CLINICAL TRIAL: NCT00912821
Title: Effect of Different Dialysis Dosage on Prognosis in Maintenance Peritoneal Dialysis Patients - A Prospective, Randomized, Controlled, Multi-center Clinical Study
Brief Title: Effect of Different Dialysis Dosage on Prognosis in Maintenance Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Aiwu Lin, Vice Director, Department of Nephrology, Renji Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08dz1900501-b
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: End-stage Renal Disease
Keywords: Renal Replacement Therapy; Peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dialysis Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 8 L dialysate (Active Comparator): 8 L peritoneal dialysis solution
  Interventions: Drug: 8 L dialysate
- 6 L dialysate (Experimental): 6 L peritoneal dialysis solution
  Interventions: Drug: 6 L dialysate

INTERVENTIONS:
Drug: 6 L dialysate — 6 L peritoneal dialysis solution
  Arms: 6 L dialysate
Drug: 8 L dialysate — 8 L peritoneal dialysis solution
  Arms: 8 L dialysate

SUMMARY:
Peritoneal dialysis (PD) is an important model of renal replacement therapy for end-stage renal disease (ESRD) patients. Thus far, evidence for the initiation dosage of PD treatment is lacking, most patients begin their PD with four 2 L exchanges per day. However, many patients have their residual renal function at the initiation of PD, an 8 L dialysate per day will enhance the toxicity of bioincompatible dialysate and increase the economic burden compared with that of 6 L dialysate per day. Thus, the investigators perform a prospective, randomized, controlled, multi-center clinical study. The patients initiation of PD treatment within 6 months are randomized to be assigned to two groups: 6 L of dialysate per day and 8 L of dialysate per day, follow up will be regularly performed until 96 weeks. Clinical outcomes such as mortality, complications and life quality between the two groups will be investigated.

DETAILED DESCRIPTION:
To investigate the effect, feasibility and safety of 6L of dialysate per day after initiation of peritoneal dialysis (PD), we perform a prospective, randomized, controlled, multi-center clinical study. The patients initiation of PD treatment within 6 months are randomized to be assigned to two groups: 6L of dialysate per day and 8L of dialysate per day, follow up will be regularly performed at baseline, 4 weeks, 8 weeks, 12 weeks, 24 weeks, 36 weeks, 48 weeks, 60 weeks, 72 weeks, 84 weeks and 96 weeks. Serum biochemical parameters, Kt/V, residual renal function (RRF), life quality and cardiovascular test will be regularly recorded. Clinical outcomes such as mortality, technique failure, complications and life quality between the two groups will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80, male or female.
2. End stage renal disease patients (eGFR < 15 ml/min/1.73 m2).
3. Maintenance peritoneal dialysis within 6 months after initiation of PD.
4. With informed consent.

Exclusion Criteria:

1. Acute renal injury.
2. Patients with an expected follow up less than 6 months sch as renal transplantation.
3. Transferred from hemodialysis or renal transplantation.
4. Residual renal function eGFR less than 1 ml/min.
5. HIV positive.
6. Cancer patients.
7. Unstable organ disease such as active tuberculosis and severe hepatitis. Patients with an expected follow up less than 48 weeks, such as planned kidney transplant.
8. Other conditions regarded as unsuitability by investigator, such as pregnancy, severe malnutrition and recent peritonitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
clinical outcome including mortality and technical failure | 2 years

SECONDARY OUTCOMES:
complications including cardiovascular disease, nutritional and inflammation status, calcium and phosphorus level, anemia and life quality | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University school of medicine, Shanghai, China